CLINICAL TRIAL: NCT01169571
Title: Phase 4, Open-Label Study Evaluating the Hemodynamic Effect of Differing Loading Regimens of Precedex in a Post-Surgical Intensive Care Patient Population
Brief Title: Study to Evaluate Hemodynamic Effect of Different Loading Doses of Precedex in Post-surgical Intensive Care Unit (ICU) Patients
Status: Completed | Type: Observational
Sponsor: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: DEX-10-03
Record Dates: First submitted 2010-07-21; First posted 2010-07-26 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Intensive Care Unit
Keywords: Initially intubated; Mechanically ventilated; Post-surgical
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group I - No loading dose: No loading dose to be administered during the loading-dose paradigms
  Interventions: Drug: Dexmedetomidine
- Group II - Loading dose over 10 minutes: Loading dose dexmedetomidine 1 mcg/kg administered over 10 minutes during the loading-dose paradigms
  Interventions: Drug: Dexmedetomidine
- Group III - Loading dose over 20 minutes: Loading dose dexmedetomidine 1 mcg/kg administered over 20 minutes during the loading-dose paradigms
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine

SUMMARY:
The objective of this study is to characterize the hemodynamic effects of Precedex (dexmedetomidine (DEX)) during 3 loading-dose paradigms in mechanically ventilated post-surgical subjects in an intensive care setting.

ELIGIBILITY:
Inclusion Criteria:

1. Subject or the subject's legally authorized representative has voluntarily signed and dated the informed consent document approved by the Research Ethics Board (REB).
2. Initially intubated and mechanically ventilated adult post-operative subjects in an intensive care setting (e.g., post operative care unit, post anesthesia care unit, etc.) that are expected to require sedation for at least 2 hours.
3. Has an American Society of Anesthesiologist (ASA) classification of 1, 2, 3 or 4.

   ASA Physical Status Classification System
   * P1 A normal healthy subject
   * P2 A subject with mild systemic disease
   * P3 A subject with severe systemic disease
   * P4 A subject with severe systemic disease that is a constant threat to life
   * P5 A moribund subject who is not expected to survive without the operation
   * P6 A declared brain-dead subject whose organs are being removed for donor purposes.
4. If female, subject must be postmenopausal, surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy), or practicing at least one of the following methods of birth control:

   * hormonal contraceptives (oral, parenteral or transdermal) for at least 3 months prior to study drug administration
   * intrauterine device (IUD)
   * double-barrier method (condoms, contraceptive sponge, diaphragm or vaginal ring with spermicidal jellies or cream).

Exclusion Criteria:

1. Subjects <18 years of age.
2. Subjects with a 2nd degree Mobitz Type II or 3rd degree heart block, unless the subject has a permanent pacemaker or pacing wires are in situ.
3. Subjects with a known allergy to dexmedetomidine.
4. Hypotension based on repeat assessments prior to (within 15 minutes) starting study drug defined as Systolic BP <90 mmHg or Diastolic BP <60 mmHg.
5. Pre-existing bradycardia prior (within 15 minutes) to starting study drug defined as HR <50 bpm.
6. Subjects who, in the opinion of the Investigator, have any other condition where the risks of dexmedetomidine would be expected to outweigh its benefits (e.g., cardiogenic shock on >2 vasopressors, death anticipated within 48 hours).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Initially intubated and mechanically ventilated post-surgical adult male and female subjects in an intensive care setting.
Sampling Method: Non-Probability Sample
Enrollment: 373 (Actual)
Dates: Start 2010-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Incidence of clinically meaningful hemodynamic abnormality (CMHA) | During the first 2 hours of study drug administration
  Clinically meaningful hemodynamic abnormalities (CMHA) consist of (any):
  * Heart Rate (HR): A native HR <40 bpm (beats per minute); HR <50 bpm requiring pharmacological intervention; systolic BP <80 mm Hg; if pacing wires are in situ, use of a pacemaker after the start of study drug.
  * Vasoactive Agent Use (i.e. vasopressor or inotrope): the need to add an additional agent to maintain BP; doubling of the dose of any vasoactive agent that was infusing at the start of the study drug.
  * Paradoxical hypertension: the need to add an additional vasodilating agent for control of hypertension; doubling of the dose of any vasodilating agent that was infusing at the start of the study drug.

SECONDARY OUTCOMES:
Incidence of clinically meaningful hemodynamic abnormality (CMHA) during the maintenance infusion period. | Maintenance infusion period (2 to 24 hours)
Incidence of adverse events (AEs) between the 3 loading-dose paradigms | Post-dexmedetomidine 24-hour observation period
  Adverse events including agitation/anxiety, cardiac dysrhythmias, rebound phenomenon, and signs of withdrawal
Incidence of paradoxical hypertension | During the first 2 hours of the post-dexmedetomidine observation period
Incidence of paradoxical hypertension | Post-dexmedetomidine 24-hour observation period
Amount of analgesics administered | 2 hours prior, and for the first 2 hours during, study drug administration
Amount of sedatives administered | 2 hours prior, and for the first 2 hours during, study drug administration

CONTACTS AND LOCATIONS:
Locations (17):
- Canada (17):
  - Foothills Medical Centre, University of Calgary, Calgary, Alberta
  - University of Alberta Hospital, Department of Anesthesiology and Pain Medicine, Edmonton, Alberta
  - Red Deer Regional Hospital Centre, Alberta Health Services, Red Deer, Alberta
  - Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Capital Health-Queen Elizabeth II Health Sciences Center, Halifax, Nova Scotia
  - Kingston General Hospital, Kingston, Ontario
  - St. Mary's General Hospital, Kitchener, Ontario
  - University Hospital, London, Ontario
  - Thunder Bay, Ontario
  - Department of Anesthesia, St. Michael's Hospital, Toronto, Ontario
  - Toronto General Hospital, University Health Network, Department of Anesthesia and Pain Management, Toronto, Ontario
  - McGill University Health Centre (MUHC) Royal Victoria Hospital (RVH), Montreal, Quebec
  - McGill University Health Centre, Montreal General Hospital (MGH), Montreal, Quebec
  - Sir Mortimer B. Davis Jewish General Hospital, Montreal, Quebec
  - Universite de Sherbrooke, Sherbrooke, Quebec
  - Département d'anesthésiologie, Institut universitaire de cardiologie et de pneumologie de Québec, Québec